CLINICAL TRIAL: NCT04568317
Title: Integration of a Smartwatch Within an Internet-delivered Intervention for Depression: a Feasibility Randomized Controlled Trial on Acceptance
Brief Title: Smartwatch-supported Internet-delivered Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silver Cloud Health (Other)
Collaborators: University of Dublin, Trinity College (Other); Berkshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20/WA0206
Record Dates: First submitted 2020-09-10; First posted 2020-09-29 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Depression
Keywords: patient acceptance; internet-delivered treatment; depression; self-monitoring; smartwatch; wearable
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Upon giving consent, participants will be randomised in two arms: iCBT intervention (n=35) and iCBT intervention with smartwatch (n=35). Participants who decline consent will be excluded from the study and will receive iCBT treatment as usual. The sample size of 70 aligns with the literature around desired sample sizes for feasibility and acceptability studies (Teare et al., 2014). Participants will be recruited regardless of whether they own a smartwatch. As the smartwatch is a new addition to the iCBT intervention, this will be the first time for all participants using a smartwatch within the 'Space from Depression' program. The degree to which participants' experience/familiarity with the smartwatch technology influenced acceptance outcomes will be investigated in a secondary analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartwatch group (Experimental): iCBT intervention 'Space from Depression' with smartwatch as an additional means to self-report data on mood, sleep and physical activity in the 'Space from Depression' program (n=35).
  Interventions: Behavioral: Space from Depression; Device: Mood Monitor watch app
- Treatment as usual group (Active Comparator): iCBT intervention 'Space from Depression' (n=35).
  Interventions: Behavioral: Space from Depression

INTERVENTIONS:
Behavioral: Space from Depression — This is a 7-module internet-based CBT program. The structure and content of the modules follow evidence-based CBT principles; they are structured to incorporate quizzes, videos, psychoeducational content and interactive tools, personalised homework suggestions and summaries. One of the interactive tools is the mood monitor, where users are encouraged to monitor their mood and reflect on several factors that might had influenced it. Clients are allocated to a psychological wellbeing practitioner (PWP). The PWP is responsible for monitoring and guiding the client's progress throughout the intervention. Over the course of the 8 week supported intervention period, on 6 separate occasions the PWP will review participants progress, leaving feedback for them and responding to the work they have completed. The basic share level allows PWP is to view users' goals for the week, key messages and progress points. Each PWP will provide post-session feedback of between 10 and 15 minutes per session.
Device: Mood Monitor watch app — The Mood Monitor watch app will allow in-the-moment self-report of patients' mood and automated monitoring of their sleep and activity level. This data will be integrated into the existing Mood Monitor tool within the participant's Space from Depression program. During the intervention, prompts to record mood data will appear on the watch app; participants will be encourage to choose the frequency and time ranges to receive prompts. The watch app main screen will provide a daily and weekly visualisation of participant's mood, bedtime, hours slept and steps count, and visual cues on their progress. Participants will receive encouragement prompts to reward frequent and consistent self-report of mood over time and a good sleep hygiene. Finally, the app "Tips to Stay Well" feature will allow participants to go through a list of lifestyle-related tips extracted from the Space from Depression program.
  Arms: Smartwatch group

SUMMARY:
The current study seeks to investigate the acceptance of the use of a smartwatch in an internet-delivered Cognitive Behavioural Therapy (CBT) based intervention for depression.

DETAILED DESCRIPTION:
Eligible patients (n=70) will be invited to use the supported intervention over an 8-week period. Participants who have indicated consent will be randomised in two arms: iCBT intervention - treatment as usual (n=35) and iCBT intervention with smartwatch (n=35). Participants in the smartwatch group will be lent a smartwatch for the duration of treatment, with an app allowing them to monitor their mood in the moment, and keep track of their daily sleep and activity level. All participants will be asked to complete an acceptance questionnaire regarding the technology at three time points: before first use, at 3 weeks, and 8 weeks. This study will contribute to the growing literature on acceptance of technology supporting mental health interventions worldwide. The results may help to establish criteria for patient acceptance of the smartwatch technology as a treatment enhancer in the context of mental health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the internet-delivered CBT intervention 'Space from Depression'
* Own a compatible mobile device (iPhone 6 or upper)

Exclusion Criteria:

* Suicidal intent/ideation; score >2 on PHQ-9 question 9
* Psychotic illness
* Alcohol or drug misuse
* Previous diagnosis of an organic mental health disorder
* Currently in psychological treatment for depression symptoms
* Unstable medication regimens

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Patient acceptance (questionnaire) | Upon consent, at 3 weeks, and at 8 weeks
  All participants will be asked to fill in the Acceptability Questionnaire (AQ) upon consent, at 3 weeks, and at 8 weeks. These measurement points are aligned with Nadal et al. (2020) Technology Acceptance Lifecycle model. The questionnaire is based on the acceptance factors identified by Kim & Park (2012). The wording of the AQ is adapted to the technology in question (smartwatch vs mobile/desktop app). Participants will rate each statement on a 5-point Likert Scale. The 8-week AQ contains a series of open-ended questions for the smartwatch group to explore additional factors that might influence the watch app acceptance (privacy protection, resistance to change, etc.).
Patient acceptance (interview) | 8 weeks
  Participants in the smartwatch group who have indicated consent in taking part in the follow-up interview will be contacted after answering the final acceptance questionnaire.
Patient acceptance (Satisfaction with Treatment measure) | Immediately after the intervention
  The SAT (Richards et al, 2013) will be used to assess patient satisfaction with the intervention. This 5-item questionnaire has been used previously to evaluate different aspects of patient satisfaction and experience with the 'Space from Depression' intervention (Richards et al, 2013).
  Score varies from 0 to 20; a higher score indicates a better outcome. The score is informed by 2 open-ended questions at the end of the questionnaire.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline - At every meeting between participant and supporter - Immediately after the intervention
  The PHQ-9 is a nine-item self-report measure of depression (Kroenke et al, 2001; Spitzer et al, 1999) that has been widely used in research and is employed as a clinical outcome measure in IAPT as part of its minimum dataset. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (A.P. Association, 2013).
  Score varies from 0 to 27; a higher score indicates a worse outcome.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline - At every meeting between participant and supporter - Immediately after the intervention
  The GAD-7 (Spitzer et al, 2006) is used nationally as a screening and outcome measure in IAPT and is part of the minimum dataset. The seven items measuring anxiety symptoms and severity reflect the DSM-Fifth Edition diagnostic criteria for GAD (A.P. Association, 2013).
  Score varies from 0 to 21; a higher score indicates a worse outcome.
Work and Social Adjustment Scale (WSAS) | Baseline - At every meeting between participant and supporter - Immediately after the intervention
  This is a five-item self-report questionnaire of functional impairment (Mundt et al, 2002) that is employed nationally as an outcome measure in IAPT. It examines the experiential impact of a disorder across different life domains from the perspective of the service users. The questionnaire examines the degree of impairment caused by a disorder on a daily basis across five dimensions: work, social life, home life, private life, and close relationships.
  Score varies from 0 to 40; a higher score indicates a worse outcome.
Usage of the program | at treatment completion, in average 8 weeks.
  Usage data in terms of time spent in the platform, number of logins, number of tools used, percentage viewed, and number of reviews will be collected. Also, the amount of mood monitor entries, sleep and activity data will be extracted. Approximate activity levels (graded 1 to 5) and sleep patterns will be analyzed to explore the changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — Silver Cloud Health; Sarah Sollesse, MSc, Principal Investigator — Berkshire Healthcare NHS Foundation Trust; Camille Nadal, MSc, Study Chair — University of Dublin, Trinity College; Gavin Doherty, PhD, Study Chair — University of Dublin, Trinity College
Locations (1):
- Berkshire Healthcare NHS Foundation Trust, Bracknell, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadal C, Earley C, Enrique A, Vigano N, Sas C, Richards D, Doherty G. Integration of a smartwatch within an internet-delivered intervention for depression: Protocol for a feasibility randomized controlled trial on acceptance. Contemp Clin Trials. 2021 Apr;103:106323. doi: 10.1016/j.cct.2021.106323. Epub 2021 Feb 20. PMID 33621632